CLINICAL TRIAL: NCT00593541
Title: Development of New Software Capabilities for Use With Cardiovascular Magnetic Resonance Imaging
Acronym: CVMRI
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator is deceased
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200210689
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Abnormalities, Cardiovascular
Keywords: MRI
MeSH Terms: conditions — Cardiovascular Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This Protocol is intended to facilitate development and testing of new cardiovascular MRI software capabilities by UC Davis Research Faculty, as well as to facilitate the evaluation of new software capabilities provided by GE and Siemens.

DETAILED DESCRIPTION:
This protocol will permit normal subjects, as well as patients with suspected or proven medical conditions, to undergo MRI studies using the new software capabilities. This Protocol is not restricted to imaging of a particular organ system or disease. The Protocol does not involve injection of any contrast agent, or other minimally-invasive or invasive procedure. It is intended only for those cases for which the only requirement of the subject is to relax and lie still while imaging is being performed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ability to give informed, written consent
* Not Pregnant or breastfeeding

Exclusion Criteria:

* Electrically, magnetically, or mechanically activated implants (for example, cardiac-pacemakers)
* Ferromagnetic implant, such as an aneurysm clip, surgical clip, or prosthesis
* History of uncontrolled claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Noraml volunteers and patients with known or suspected cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 1999-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Extend or generalize certain capabilities, such as new data acquisition pulse sequences, new image processing and analysis software for structural and functional analysis of the MR images | Post-scanning

SECONDARY OUTCOMES:
Improve image quality by various techniques (e.g. reducing the effects of motion) | Post-scanning

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Buonocore, MD, PhD, Principal Investigator — University of California, Davis